CLINICAL TRIAL: NCT00643760
Title: Study PXN110448: A Dose-response Study of XP13512, Compared With Concurrent Placebo Control and LYRICA(Pregabalin), in Subjects With Neuropathic Pain Associated Withdiabetic Peripheral Neuropathy (DPN)
Brief Title: A Study In Patients With Neuropathic Pain From Diabetic Peripheral Neuropathy (DPN)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: XenoPort, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 110448
Record Dates: First submitted 2008-02-19; First posted 2008-03-26 (Estimated); Results first posted 2011-05-11 (Estimated); Last update posted 2013-07-22 (Estimated); Status verified 2013-01

CONDITIONS: Neuropathy, Diabetic
Keywords: Peripheral Diabetic Neuropathy (PDN); Neuropathic Pain
MeSH Terms: conditions — Diabetic Neuropathies; Neuralgia | interventions — 1-(((alpha-isobutanoyloxyethoxy)carbonyl)aminomethyl)-1-cyclohexaneacetic acid; Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Pregabalin (Other): Pregabalin 300mg/day (positive control), maintenance treatment 14 weeks
  Interventions: Drug: Pregabalin
- GEn 1200mg/day (Experimental): gabapentin enacarbil 1200mg/day, maintenance treatment 14 weeks
  Interventions: Drug: GEn 1200mg/day
- GEn 2400mg/day (Experimental): gabapentin enacarbil 2400mg/day, maintenance treatment 14 weeks
  Interventions: Drug: GEn 2400mg/day
- GEn 3600mg/day (Experimental): gabapentin enacarbil 3600mg/day, maintanance treatment 14 weeks
  Interventions: Drug: GEn 3600mg/day

INTERVENTIONS:
Drug: Placebo — placebo
  Arms: Placebo
Drug: GEn 1200mg/day — gabapentin enacarbil 1200mg/day
  Other Names: XP13512; GSK1838262; gabapentin enacarbil
  Arms: GEn 1200mg/day
Drug: GEn 2400mg/day — gabapentin enacarbil 2400mg/day
  Other Names: gabapentin enacarbil; GSK1838262; XP13512
  Arms: GEn 2400mg/day
Drug: GEn 3600mg/day — gabapentin enacarbil 3600mg/day
  Other Names: XP13512; GSK1838262; gabapentin enacarbil
  Arms: GEn 3600mg/day
Drug: Pregabalin — pregabalin 300mg/day
  Arms: Pregabalin

SUMMARY:
The purpose of this study is to determine whether gabapentin enacarbil (XP13512/GSK1838262), hereafter referred to as GEn is effective in the treatment of neuropathic pain associated with diabetic peripheral neuropathy(DPN)

DETAILED DESCRIPTION:
This is a dose-response study of XP13512 compared with concurrent placebo control and LYRICA (pregabalin), in subjects with neuropathic pain associated with DPN. Three doses of XP13512 (1200 mg/day, 2400 mg/day and 3600 mg/day) are being evaluated for the management of neuropathic pain associated with DPN. Approximately 392 subjects from 70 to 80 participating sites in the US will be randomized to receive either XP13512 at the above mentioned doses, placebo or pregabalin (300mg/day).

ELIGIBILITY:
Inclusion criteria:

* 18 years or older
* Female subjects are eligible to enter if of non-childbearing potential or not lactating, has a negative pregnancy test and agrees to use a specified highly effective method for avoiding pregnancy
* Documented medical diagnosis of Type 1 or 2 diabetes including:
* Stable glycemic control for 3 months defined as <25% change of routine insulin, <50% change of routine oral anti-diabetic agent dose and HbA1c < 8%. (HbA1c of 8 to 11% eligible if attempts to improve diabetic control failed)
* DPN defined by:
* Bilateral reduced or absent reflexes at the ankles, or
* Bilateral impaired vibration, pinprick, fine touch or temperature perception in the distal lower extremities And
* Persistent distal burning or dull pain in the feet, or
* Persistent proximal aching pain in the legs, or
* Paroxysmal electric, shooting, stabbing pain, or
* Dysasthesias, or
* Evoked pain And
* history of pain for at least six months and no greater than five years attributed to DPN (refers to duration of pain)
* Baseline 24-hour average daily pain intensity score >4.0 as measured on an 11 point pain intensity numerical rating scale
* Provides written informed consent in accordance with all applicable regulatory requirements

Exclusion criteria:

* Other chronic pain conditions not associated with DPN. However, the subject will not be excluded if:
* The pain condition is located at a different region of the body, and
* The pain intensity of this condition is not greater than the pain intensity of the DPN, and
* The subject can assess their DPN independently of other pain condition.
* Other causes of neuropathy or lower extremity pain
* Is unable to discontinue prohibited medications or non-drug therapies or procedures throughout the duration of the study
* Hepatic impairment defined as ALT or AST > 2x upper limit of normal (ULN) or alkaline phosphatase or bilirubin > 1.5x ULN
* Chronic hepatitis B or C
* Impaired renal function defined as either creatinine clearance < 60 mL/min or requiring hemodialysis
* Corrected QT (QTc) interval >450 msec or QTc interval >480 msec for patients with Bundle Branch Block
* Uncontrolled hypertension at screen (sitting systolic >160 mmHg and/or sitting diastolic >90 mmHg
* Current diagnosis of active epilepsy or any active seizure disorder requiring chronic therapy with antiepileptic drug(s)
* Medical condition or disorder that would interfere with the action, absorption, distribution, metabolism, or excretion of GEn or pregabalin, or, in the investigator's judgment:
* Is considered to be clinically significant and could pose a safety concern or,
* Could interfere with the accurate assessment of safety or efficacy, or,
* Could potentially affect a subject's safety or study outcome
* Meets criteria defined by the DSM-IV-TR for a major depressive episode or for active significant psychiatric disorders within last year
* Depression in remission, with or without antidepressant treatment, may participate, unless stable antidepressant regimen is a prohibited medication
* Antidepressant medication may not be changed or discontinued to met entry criteria and must be stable for at least 3 months prior to enrollment
* History of clinically significant drug or alcohol abuse (DSM-IV-TR). Benzodiazepines or atypical benzodiazepines as hypnotic sleep agents permitted
* Currently participating in another clinical study in which the subject is, or will be exposed to an investigational or non-investigational drug or device
* Has participated in a clinical study and was exposed to investigational or non-investigational drug or device:
* Within preceding month for studies unrelated to DPN, or
* Within six months for studies related to DPN
* Treated previously with GEn
* History of allergic or medically significant adverse reaction to investigational products (including gabapentin or pregabalin) or their excipients, acetaminophen or related compounds

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 421 (Actual)
Dates: Start 2008-03; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (84):
- United States (84):
  - GSK Investigational Site, Alabaster, Alabama
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Dothan, Alabama
  - GSK Investigational Site, Hoover, Alabama
  - GSK Investigational Site, Jasper, Alabama
  - GSK Investigational Site, Muscle Shoals, Alabama
  - GSK Investigational Site, Northport, Alabama
  - GSK Investigational Site, Tuscaloosa, Alabama
  - GSK Investigational Site, Mesa, Arizona
  - GSK Investigational Site, Peoria, Arizona
  - GSK Investigational Site, Tempe, Arizona
  - GSK Investigational Site, Hot Springs, Arkansas
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Anaheim, California
  - GSK Investigational Site, Concord, California
  - GSK Investigational Site, Escondido, California
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Huntington Park, California
  - GSK Investigational Site, La Jolla, California
  - GSK Investigational Site, Los Gatos, California
  - GSK Investigational Site, Mission Viejo, California
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, Northridge, California
  - GSK Investigational Site, Oxnard, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Santa Ana, California
  - GSK Investigational Site, Santa Monica, California
  - GSK Investigational Site, Temecula, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, Westlake Village, California
  - GSK Investigational Site, Brandon, Florida
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Fort Myers, Florida
  - GSK Investigational Site, Hallandale, Florida
  - GSK Investigational Site, Hollywood, Florida
  - GSK Investigational Site, New Port Richey, Florida
  - GSK Investigational Site, Ocala, Florida
  - GSK Investigational Site, Ormond Beach, Florida
  - GSK Investigational Site, Pembroke Pines, Florida
  - GSK Investigational Site, St. Petersburg, Florida
  - GSK Investigational Site, Tallahassee, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Marietta, Georgia
  - GSK Investigational Site, Roswell, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Libertyville, Illinois
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Rockville, Maryland
  - GSK Investigational Site, Wellesley Hills, Massachusetts
  - GSK Investigational Site, Kalamazoo, Michigan
  - GSK Investigational Site, Olive Branch, Mississippi
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Flushing, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, North Massapequa, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Staten Island, New York
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Salisbury, North Carolina
  - GSK Investigational Site, Toledo, Ohio
  - GSK Investigational Site, Norman, Oklahoma
  - GSK Investigational Site, Eugene, Oregon
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Levittown, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Greer, South Carolina
  - GSK Investigational Site, Mt. Pleasant, South Carolina
  - GSK Investigational Site, Kingsport, Tennessee
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Alexandria, Virginia
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Weber City, Virginia
  - GSK Investigational Site, Spokane, Washington
  - GSK Investigational Site, Tacoma, Washington
  - GSK Investigational Site, Vancouver, Washington

REFERENCES:
- [Derived] Rauck R, Makumi CW, Schwartz S, Graff O, Meno-Tetang G, Bell CF, Kavanagh ST, McClung CL. A randomized, controlled trial of gabapentin enacarbil in subjects with neuropathic pain associated with diabetic peripheral neuropathy. Pain Pract. 2013 Jul;13(6):485-96. doi: 10.1111/papr.12014. Epub 2012 Nov 27. PMID 23186035

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Three 600 milligram (mg) gabapentin enacarbil (XP13512/GSK1838262), hereafter referred to as GEn, placebo tablets taken orally twice daily (morning and evening); one 100 mg pregabalin (PGB) placebo capsule taken orally three times daily (morning, midday, and evening).
- GEn 1200 mg/Day: One 600 mg extended release (ER) GEn tablet and two 600 mg GEn placebo tablets taken orally twice daily (morning and evening); one 100 mg PGB placebo capsule taken orally three times daily (morning, midday, and evening).
- GEn 2400 mg/Day: Two 600 mg ER GEn tablets and one 600 mg GEn placebo tablet taken orally twice daily (morning and evening); one 100 mg PGB placebo capsule taken orally three times daily (morning, midday, and evening).
- GEn 3600 mg/Day: Three 600 mg ER GEn tablets taken orally twice daily (morning and evening); one 100 mg PGB placebo capsule taken orally three times daily (morning, midday, and evening).
- PGB 300 mg/Day: Three 600 mg GEn placebo tablets taken orally twice daily (morning and evening); one 100 mg PGB capsule taken orally three times daily (morning, midday, and evening).
Period: Overall Study
Arm/Group | Placebo | GEn 1200 mg/Day | GEn 2400 mg/Day | GEn 3600 mg/Day | PGB 300 mg/Day
Started | 120 | 62 | 56 | 117 | 66
Safety Population/Treated With Drug | 120 | 62 | 56 | 116 | 66
ITT Population | 120 | 62 | 56 | 116 | 66
Completed | 90 | 47 | 37 | 79 | 47
Not Completed | 30 | 15 | 19 | 38 | 19
Not completed — Adverse Event | 11 | 5 | 12 | 21 | 6
Not completed — Lack of Efficacy | 3 | 1 | 0 | 4 | 3
Not completed — Protocol Violation | 7 | 6 | 4 | 4 | 6
Not completed — Lost to Follow-up | 6 | 2 | 1 | 3 | 3
Not completed — Investigator Discretion | 0 | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 2 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | GEn 1200 mg/Day | GEn 2400 mg/Day | GEn 3600 mg/Day | PGB 300 mg/Day | Total
Number analyzed (Participants) | 120 | 62 | 56 | 116 | 66 | 420
Age Continuous [Mean (Standard Deviation); unit: Years] — Age in years of the Intent-to-Treat (ITT) Population, comprised of all randomized participants who took at least one dose of investigational product and provided at least one post-baseline efficacy measurement, was used for all baseline characteristics. This population does not include all participants randomized to study treatment.
  Years | 60.1 (10.63) | 57.5 (10.32) | 60.8 (8.97) | 57.5 (9.87) | 57.7 (10.59) | 58.7 (10.20)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender of the ITT Population, comprised of all randomized participants who took at least one dose of investigational product and provided at least one post-baseline efficacy measurement, was used for all baseline characteristics. This population does not include all participants randomized to study treatment.
  Participants
    Female | 47 | 28 | 19 | 45 | 32 | 171
    Male | 73 | 34 | 37 | 71 | 34 | 249
Race/Ethnicity, Customized [Number; unit: participants] — Race of the ITT Population, comprised of all randomized participants who took at least one dose of investigational product and provided at least one post-baseline efficacy measurement, was used for all baseline characteristics. This population does not include all participants randomized to study treatment.
  participants
    African American/African Heritage | 20 | 15 | 7 | 20 | 12 | 74
    American Indian or Alaskan Native | 2 | 0 | 0 | 0 | 0 | 2
    Asian - Central/South Asian Heritage | 0 | 0 | 0 | 1 | 0 | 1
    Asian - South East Asian Heritage | 0 | 1 | 0 | 2 | 0 | 3
    White - Arabic/North African Heritage | 0 | 2 | 2 | 1 | 0 | 5
    White - White/Caucasian/European Heritage | 98 | 44 | 45 | 89 | 52 | 328
    Mixed Race | 0 | 0 | 1 | 1 | 0 | 2
    Not Provided | 0 | 0 | 1 | 2 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Mean 24-hour Average Pain Intensity (API) Score at End of Maintenance Treatment (EOMT) Using Last Observation Carried Forward (LOCF) Data
Description: Baseline and EOMT values are the calculated means of the daily 24-hour API scores for each participant during the last 7 days prior to randomization (Baseline) and the earliest date of Week 13 visit/Withdrawal visit/last dose of study drug (EOMT). Participants used a hand-held diary to rate their API over the preceding 24 hours, using an 11-point Pain Intensity Numerical Rating Scale (PI-NRS) (0=no pain, 10=pain as bad as you can imagine). LOCF was used if less than 4 days of diary data were provided. Change from baseline was calculated as the EOMT score minus the Baseline score.
Time Frame: Baseline and EOMT (representing the earliest date of Week 13 visit/withdrawal visit)
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | GEn 1200 mg/Day | GEn 2400 mg/Day | GEn 3600 mg/Day | PGB 300 mg/Day
Number analyzed (Participants) | 120 | 62 | 56 | 116 | 66
scores on a scale | -2.08 (0.196) | -2.43 (0.274) | -2.10 (0.289) | -2.63 (0.202) | -1.65 (0.266)
Statistical Analysis 1: Comparison: Placebo vs GEn 1200 mg/Day; Test type: Superiority or Other; p = 0.295, ANCOVA — This p-value has been adjusted for multiplicity using a combination of a sequential method and the Hochberg procedure in order to maintain the overall experiment-wise alpha level of 0.05; Analysis of covariance (ANCOVA) model with body mass index (BMI), baseline 24-hour average pain intensity, and grouped center as covariates was used; Adjusted mean difference versus placebo = -0.35, 95% CI [-1.02 to 0.31]
Statistical Analysis 2: Comparison: Placebo vs GEn 2400 mg/Day; Test type: Superiority or Other; p = 0.946, ANCOVA — [p-value comment as in outcome 1, analysis 1]; An ANCOVA model with BMI, baseline 24-hour average pain intensity, and grouped center as covariates was used; Adjusted mean difference versus placebo = -0.02, 95% CI [-0.71 to 0.66]
Statistical Analysis 3: Comparison: Placebo vs GEn 3600 mg/Day; Test type: Superiority or Other; p = 0.105, ANCOVA — [p-value comment as in outcome 1, analysis 1]; An ANCOVA model with BMI, baseline 24-hour average pain intensity, and grouped center as covariates was used; Adjusted mean difference versus placebo = -0.55, 95% CI [-1.10 to 0.01]
Statistical Analysis 4: Comparison: Placebo vs PGB 300 mg/Day; Test type: Superiority or Other; Adjusted mean difference versus placebo = 0.43, 95% CI [-0.22 to 1.08]

2. Secondary Outcome: Change From Baseline in the Mean Day-time Average Pain Intensity (API) Score at EOMT Using LOCF Data
Description: Day-time is defined as the time between rising in the morning and going to bed at night. Participants recorded day-time API on a daily basis in the evening before bedtime using an 11-point PI-NRS (0=no pain, 10=pain as bad as you can imagine). Baseline and EOMT are as defined for the primary endpoint. Change from baseline was calculated as the EOMT score minus the baseline score. An ANCOVA model with baseline value, BMI, grouped center as covariates was used.
Time Frame: Baseline and EOMT (representing the earliest date of Week 13 visit/withdrawal visit)
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | GEn 1200 mg/Day | GEn 2400 mg/Day | GEn 3600 mg/Day | PGB 300 mg/Day
Number analyzed (Participants) | 120 | 62 | 56 | 116 | 66
scores on a scale | -2.07 (0.195) | -2.35 (0.272) | -2.06 (0.286) | -2.54 (0.200) | -1.50 (0.264)

3. Secondary Outcome: Change From Baseline in the Mean Night-time Average Pain Intensity (API) Score at EOMT Using LOCF Data
Description: Night-time is defined as the time between going to bed at night and rising in the morning. Participants recorded night-time API on a daily basis in the morning upon awakening using an 11-point PI-NRS (0=no pain, 10=pain as bad as you can imagine). Baseline and EOMT are as defined for the primary endpoint. Change from baseline was calculated as the EOMT score minus the baseline score. An ANCOVA model with baseline value, BMI, grouped center as covariates was used.
Time Frame: Baseline and EOMT (representing the earliest date of Week 13 visit/withdrawal visit)
Population: ITT Population. There were two participants in the GEn 3600 mg/day group who did not complete enough post-baseline morning diaries to calculate an average night-time pain intensity score for the EOMT timepoint.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | GEn 1200 mg/Day | GEn 2400 mg/Day | GEn 3600 mg/Day | PGB 300 mg/Day
Number analyzed (Participants) | 120 | 62 | 56 | 114 | 66
scores on a scale | -1.99 (0.203) | -2.15 (0.282) | -2.04 (0.298) | -2.71 (0.210) | -1.83 (0.274)

4. Secondary Outcome: Change From Baseline in the Mean Current (Morning) Pain Intensity Score at EOMT Using LOCF Data
Description: Current pain is defined as the participant's assessment of pain intensity "right now." Participants recorded their current morning pain intensity in the morning upon wakening using an 11-point PI-NRS (0=no pain, 10=pain as bad as you can imagine). Baseline and EOMT are as defined for the primary endpoint. Change from baseline was calculated as the EOMT score minus the baseline score. An ANCOVA model with baseline value, BMI, grouped center as covariates was used.
Time Frame: Baseline and EOMT (representing the earliest date of Week 13 visit/withdrawal visit)
Population: ITT Population. There were two participants in the GEn 3600 mg/day group who did not complete enough post-baseline morning diaries to calculate a current (morning) pain intensity score for the EOMT timepoint.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | GEn 1200 mg/Day | GEn 2400 mg/Day | GEn 3600 mg/Day | PGB 300 mg/Day
Number analyzed (Participants) | 120 | 62 | 56 | 114 | 66
scores on a scale | -1.90 (0.192) | -2.08 (0.268) | -1.95 (0.282) | -2.40 (0.199) | -1.50 (0.260)

5. Secondary Outcome: Change From Baseline in the Mean Current (Evening) Pain Intensity Score at EOMT Using LOCF Data
Description: Current pain is defined as the participant's assessment of pain intensity "right now." Participants recorded their current evening pain intensity in the evening before bedtime using an 11-point PI-NRS (0=no pain, 10=pain as bad as you can imagine). Baseline and EOMT are as defined for the primary endpoint. Change from baseline was calculated as the EOMT score minus the baseline score. An ANCOVA model with baseline value, BMI, grouped center as covariates was used.
Time Frame: Baseline and EOMT (representing the earliest date of Week 13 visit/withdrawal visit)
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | GEn 1200 mg/Day | GEn 2400 mg/Day | GEn 3600 mg/Day | PGB 300 mg/Day
Number analyzed (Participants) | 120 | 62 | 56 | 116 | 66
scores on a scale | -2.19 (0.194) | -2.24 (0.271) | -2.10 (0.285) | -2.66 (0.200) | -1.65 (0.264)

6. Secondary Outcome: Change From Baseline in the Mean Day-time Worst Pain Intensity Score at EOMT Using LOCF Data
Description: Day-time worst pain is defined as the partipant's assessment of their worst pain between rising in the morning and going to bed at night. Participants recorded day-time worst pain in the evening before bedtime using an 11-point PI-NRS (0=no pain, 10=pain as bad as you can imagine). Baseline and EOMT are as defined for the primary endpoint. Change from baseline was calculated as the EOMT score minus the baseline score. An ANCOVA model with baseline value, BMI, grouped center as covariates was used.
Time Frame: Baseline and EOMT (representing the earliest date of Week 13 visit/withdrawal visit)
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | GEn 1200 mg/Day | GEn 2400 mg/Day | GEn 3600 mg/Day | PGB 300 mg/Day
Number analyzed (Participants) | 120 | 62 | 56 | 116 | 66
scores on a scale | -2.33 (0.210) | -2.35 (0.292) | -2.25 (0.307) | -2.88 (0.215) | -1.62 (0.284)

7. Secondary Outcome: Change From Baseline in the Mean Night-time Worst Pain Intensity Score at EOMT Using LOCF Data
Description: Night-time worst pain is defined as the partipant's assessment of their worst pain between going to bed at night and rising in the morning. Participants recorded night-time worst pain in the morning upon awakening using an 11-point PI-NRS (0=no pain, 10=pain as bad as you can imagine). Baseline and EOMT are as defined for the primary endpoint. Change from baseline was calculated as the EOMT score minus the baseline score. An ANCOVA model with baseline value, BMI, grouped center as covariates was used.
Time Frame: Baseline and EOMT (representing the earliest date of Week 13 visit/withdrawal visit)
Population: ITT Population. There were two participants in the GEn 3600 mg/day group who did not complete enough post-baseline morning diaries to calculate a night-time worst pain intensity score for the EOMT timepoint.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | GEn 1200 mg/Day | GEn 2400 mg/Day | GEn 3600 mg/Day | PGB 300 mg/Day
Number analyzed (Participants) | 120 | 62 | 56 | 114 | 66
scores on a scale | -2.25 (0.213) | -2.24 (0.297) | -2.25 (0.313) | -3.00 (0.221) | -1.86 (0.289)

8. Secondary Outcome: Change From Baseline in the Mean Sleep Interference Score at EOMT Using LOCF Data
Description: Participants assessed sleep interference due to pain on a daily basis in the morning upon awakening using an 11-point NRS (0=pain does not interfere with sleep, 10=pain completely interferes with sleep). Baseline and EOMT are as defined for the primary endpoint. Change from baseline was calculated as the EOMT score minus the baseline score. An ANCOVA model with baseline value, BMI, grouped center as covariates was used.
Time Frame: Baseline and EOMT (representing the earliest date of Week 13 visit/withdrawal visit)
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | GEn 1200 mg/Day | GEn 2400 mg/Day | GEn 3600 mg/Day | PGB 300 mg/Day
Number analyzed (Participants) | 120 | 62 | 56 | 114 | 66
scores on a scale | -2.35 (0.214) | -2.54 (0.298) | -2.45 (0.313) | -3.01 (0.221) | -2.24 (0.289)

9. Secondary Outcome: Change From Baseline in the Mean Daily Dose of Rescue Medication at EOMT Using LOCF Data
Description: Mean daily use of rescue medication (milligrams of acetaminophen) was calculated by determining the average number of tablets taken per day of rescue medication (Commerical Tylenol) during treatment and multiplying that by 500 mg. Baseline and EOMT are as defined for the primary endpoint. Change from baseline was calculated as the EOMT score minus the baseline score. An ANCOVA model with baseline value, BMI, grouped center as covariates was used.
Time Frame: Baseline and EOMT (representing the earliest date of Week 13 visit/withdrawal visit)
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: milligrams
Arm/Group | Placebo | GEn 1200 mg/Day | GEn 2400 mg/Day | GEn 3600 mg/Day | PGB 300 mg/Day
Number analyzed (Participants) | 120 | 62 | 56 | 116 | 66
milligrams | -261.99 (73.630) | -171.64 (102.482) | -102.51 (107.918) | -228.54 (76.139) | -246.07 (99.758)

10. Secondary Outcome: Change From Baseline in Pain Quality as Assessed by the Neuropathic Pain Scale (NPS) Summary Scores at EOMT Using LOCF Data
Description: The NPS assesses pain qualities and consists of 11-items, 10 assessed on an 11-point NRS (0=no impact to 10=greatest impact); and 1 open-ended question not used in score calculation. 4 summary scores are calculated: NPS 10 (items 1-7, 9-11), NPS 8 (8 pain descriptor items), NPS Non-Allodynic (NA) (8 NA items), and NPS 4 (4 pain quality items); and range from 0 to 100 (0=no impact and 100=greatest impact). The analysis is based on the change from baseline (BL) (EOMT score minus the BL score) using an ANCOVA model with BL value, BMI, grouped center as covariates.
Time Frame: Baseline and EOMT (representing the earliest date of Week 13 visit/withdrawal visit)
Population: ITT Population. Not all participants completed an NPS assessment at both Baseline and Week 13/Withdrawal; as such, the number analyzed is different from the full ITT Population counts.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | GEn 1200 mg/Day | GEn 2400 mg/Day | GEn 3600 mg/Day | PGB 300 mg/Day
Number analyzed (Participants) | 112 | 58 | 45 | 108 | 62
scores on a scale
  NPS 10 Score | -18.92 (1.914) | -18.43 (2.658) | -22.24 (3.027) | -25.49 (1.970) | -16.16 (2.576)
  NPS 8 Score | -18.73 (1.898) | -17.83 (2.637) | -21.84 (3.003) | -25.14 (1.954) | -16.19 (2.555)
  NPS Non-Allodynic Score | -19.37 (1.998) | -18.89 (2.776) | -22.86 (3.160) | -26.35 (2.057) | -15.63 (2.690)
  NPS 4 Score | -20.54 (2.120) | -20.90 (2.944) | -25.15 (3.352) | -27.84 (2.182) | -16.06 (2.853)

11. Secondary Outcome: Change From Baseline in Pain Characteristics and Intensity as Assessed by the Short Form-McGill Pain Questionnaire (SF-MPQ) at EOMT Using LOCF Data
Description: The SF-MPQ, a general pain instrument, assesses the characteristics and intensity of pain and consists of 15-items assessed on a 4-point scale (0=none, 1=mild, 2=moderate, and 3=severe). 3 summary scores are calculated: sensory score (sum of items 1-11, range 0-33), affective score (sum of items 12-15, range 0-12), total score (sum of items 1-15, range 0-45), where lower scores = lower pain/impact. Analysis is based on the change from baseline (BL) (EOMT score minus the BL score) using an ANCOVA model with BL value, BMI, grouped center as covariates.
Time Frame: Baseline and EOMT (representing the earliest date of Week 13 visit/withdrawal visit)
Population: ITT Population. Not all participants completed an SF-MPQ assessment at both Baseline and Week 13/Withdrawal; as such, the number analyzed is different from the full ITT Population counts.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | GEn 1200 mg/Day | GEn 2400 mg/Day | GEn 3600 mg/Day | PGB 300 mg/Day
Number analyzed (Participants) | 112 | 57 | 44 | 108 | 62
scores on a scale
  SF-MPQ Total Score | -5.85 (0.865) | -6.55 (1.214) | -6.75 (1.381) | -7.56 (0.888) | -4.01 (1.161)
  SF-MPQ Sensory Score | -4.25 (0.674) | -4.83 (0.946) | -5.31 (1.077) | -5.50 (0.692) | -2.73 (0.906)
  SF-MPQ Affective Score | -1.63 (0.247) | -1.65 (0.348) | -1.45 (0.395) | -2.07 (0.254) | -1.26 (0.332)

12. Secondary Outcome: Change From Baseline in Pain Score After Taking a 50-foot Walk at EOMT
Description: Baseline and EOMT scores are the pain scores each participant reported after taking a 50-foot walk at the randomization and Week 13/Withdrawal visits, respectively, using an 11-point PI-NRS (0=no pain, 10=pain as bad as you can imagine). Change from baseline was calculated as the EOMT score minus the baseline score. An ANCOVA model with BMI, baseline pain intensity after 50-foot walk, pain intensity prior to 50-foot walk at the visit being assessed, and grouped center as covariates was used.
Time Frame: Baseline and EOMT (representing the earliest date of Week 13 visit/withdrawal visit)
Population: ITT Population. Not all participants completed a 50-foot walk at both Baseline and Week 13/Withdrawal; as such, the number analyzed is different from the full ITT Population counts.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | GEn 1200 mg/Day | GEn 2400 mg/Day | GEn 3600 mg/Day | PGB 300 mg/Day
Number analyzed (Participants) | 111 | 57 | 44 | 107 | 59
scores on a scale | -2.38 (0.077) | -2.32 (0.107) | -2.36 (0.122) | -2.52 (0.080) | -2.17 (0.106)

13. Secondary Outcome: Number of Participants Who Are Responders on the Patient Global Impression of Change (PGIC) Questionnaire at EOMT Using LOCF Data
Description: The PGIC is a single-item questionnaire designed to provide an overall assessment of treatment from the participant's perspective since the start of the study. It is measured on a 7-point scale, where 1=very much improved and 7=very much worse. A participant is considered a responder if they have a response of "very much improved" or "much improved." EOMT response is defined as the score recorded at the Week 13/Withdrawal visit.
Time Frame: EOMT (representing the earliest date of Week 13 visit/withdrawal visit)
Population: ITT Population. Not all participants completed a PGIC assessment at Week 13/Withdrawal; as such, the number analyzed is different from the full ITT Population counts.
Measure: Number; unit: participants
Arm/Group | Placebo | GEn 1200 mg/Day | GEn 2400 mg/Day | GEn 3600 mg/Day | PGB 300 mg/Day
Number analyzed (Participants) | 112 | 58 | 46 | 108 | 62
participants | 46 | 22 | 24 | 53 | 62

14. Secondary Outcome: Number of Participants Who Are Responders on the Clinician Global Impression of Change (CGIC) Questionnaire at EOMT Using LOCF Data
Description: The CGIC is a single-item questionnaire designed to provide an overall assessment of treatment from the clinician's perspective since the start of the study. It is measured on a 7-point scale, where 1=very much improved and 7=very much worse. A participant is considered a responder if they have a response of "very much improved" or "much improved." EOMT response is defined as the score recorded at the Week 13/Withdrawal visit.
Time Frame: EOMT (representing the earliest date of Week 13 visit/withdrawal visit)
Population: ITT Population. Not all participants had a CGIC assessment at Week 13/Withdrawal; as such, the number analyzed is different from the full ITT Population counts.
Measure: Number; unit: participants
Arm/Group | Placebo | GEn 1200 mg/Day | GEn 2400 mg/Day | GEn 3600 mg/Day | PGB 300 mg/Day
Number analyzed (Participants) | 98 | 52 | 40 | 89 | 54
participants | 39 | 20 | 22 | 50 | 17

15. Secondary Outcome: Number of Participants Achieving Various Levels of Percent Reduction From Baseline in the Mean 24-hour Average Pain Intensity Score at EOMT Using LOCF Data
Description: Baseline and EOMT scores are the calculated means of the 24-hour average pain scores for each participant during the last 7 days prior to randomization and EOMT, respectively. Percent reduction from baseline was calculated as the [(EOMT score minus the baseline score)divided by the baseline score], multiplied by 100. The PI-NRS is an 11-point scale (0=no pain, 10=pain as bad as you can imagine) by which a participant assesses their 24-hour average pain intensity.
Time Frame: Baseline and EOMT (representing the earliest date of Week 13 visit/withdrawal visit)
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Placebo | GEn 1200 mg/Day | GEn 2400 mg/Day | GEn 3600 mg/Day | PGB 300 mg/Day
Number analyzed (Participants) | 120 | 62 | 56 | 116 | 66
participants
  >= 0% reduction from baseline | 103 | 55 | 50 | 101 | 55
  >= 10% reduction from baseline | 86 | 43 | 42 | 91 | 42
  >= 20% reduction from baseline | 73 | 36 | 34 | 78 | 36
  >= 30% reduction from baseline | 57 | 31 | 25 | 66 | 28
  >= 40% reduction from baseline | 46 | 28 | 19 | 55 | 20
  >= 50% reduction from baseline | 35 | 26 | 15 | 46 | 14
  >= 60% reduction from baseline | 26 | 21 | 11 | 41 | 9
  >= 70% reduction from baseline | 15 | 17 | 6 | 25 | 5
  >= 80% reduction from baseline | 11 | 11 | 5 | 17 | 4
  >= 90% reduction from baseline | 4 | 5 | 2 | 8 | 3
  100% reduction from baseline | 3 | 4 | 1 | 5 | 3

16. Secondary Outcome: Time to Onset of Sustained Improvement in the 24-hour Average Pain Intensity Score
Description: Sustained improvement in the 24-hour average pain intensity score is defined as at least 2 consecutive days on which the 24-hour average pain intensity score is >=2 points less than the mean 24-hour average pain intensity score at baseline. Time to onset is measured from baseline and was calculated as first day of event minus last day of baseline and is expressed in days. Baseline score is the calculated mean of the 24-hour average pain score for each participant during the last 7 days prior to randomization.
Time Frame: Any time post-baseline until date of last dose of study medication (up to Week 13)
Population: ITT Population
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | GEn 1200 mg/Day | GEn 2400 mg/Day | GEn 3600 mg/Day | PGB 300 mg/Day
Number analyzed (Participants) | 120 | 62 | 56 | 116 | 66
days | 24 [2 to 97] | 25 [2 to 76] | 22 [2 to 62] | 15 [1 to 87] | 29 [2 to 93]

17. Secondary Outcome: Change From Baseline in Severity of Pain and the Impact of Pain as Assessed by the Brief Pain Inventory (BPI) at EOMT Using LOCF Data
Description: The BPI, a general pain instrument, assesses the severity and interference of pain; and consists of 6 items assessed on an 11-point NRS (0=no impact and 10=greatest impact). 2 summary scores are calculated: BPI Severity Score (average of first 4 items) and BPI Interference Score (average of 7 responses to item 6); where each summary score ranges from 0 to 10 (0=no impact and 10=greatest impact). Analysis of this endpoint is based on the change from baseline (BL) (EOMT score minus the BL score) using an ANCOVA model with BL value, BMI, grouped center as covariates.
Time Frame: Baseline and EOMT
Population: ITT Population. Not all participants completed a BPI assessment at both Baseline and Week 13/Withdrawal; as such, the number analyzed is different from the full ITT Population counts.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | GEn 1200 mg/Day | GEn 2400 mg/Day | GEn 3600 mg/Day | PGB 300 mg/Day
Number analyzed (Participants) | 112 | 57 | 44 | 107 | 62
scores on a scale
  Brief Pain Inventory Severity of Pain | -2.1 (0.21) | -2.3 (0.29) | -2.4 (0.33) | -2.8 (0.21) | -1.7 (0.28)
  Brief Pain Inventory Interference of Pain | -2.0 (0.21) | -2.0 (0.30) | -2.1 (0.34) | -2.5 (0.22) | -1.9 (0.29)

18. Secondary Outcome: Change From Baseline in Quality of Life as Assessed by the 36-Item Short Form Health Survey (SF-36) at EOMT Using LOCF Data
Description: The SF-36 is a general health-related quality of life instrument consisting of 36 items with various response options (Yes/No, 5- to 6-point Likert scale). Summary scores are calculated for 8 domains and 2 components (physical and mental); where scores range from 0 to 100 (higher scores = better quality of life). Analysis of this endpoint is based on the change from baseline (BL) (EOMT score minus the BL score) using an ANCOVA model with BL value, BMI, grouped center as covariates.
Time Frame: Baseline and EOMT (representing the earliest date of Week 13 visit/withdrawal visit)
Population: ITT Population. Not all participants completed an SF-36 at both Baseline and Week 13/Withdrawal; as such, the number analyzed is different from the full ITT Population counts.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | GEn 1200 mg/Day | GEn 2400 mg/Day | GEn 3600 mg/Day | PGB 300 mg/Day
Number analyzed (Participants) | 112 | 57 | 44 | 107 | 61
scores on a scale
  SF-36 Physical Component Summary Score | 3.1 (0.67) | 3.5 (0.93) | 3.7 (1.06) | 4.6 (0.69) | 3.7 (0.90)
  SF-36 Mental Component Summary Score | 2.5 (0.88) | 0.4 (1.24) | 1.5 (1.41) | 1.6 (0.91) | 0.7 (1.20)

19. Secondary Outcome: Change From Baseline in Emotional Functioning as Assessed by the Profile of Mood States-Brief Form (POMS-B) at EOMT Using LOCF Data
Description: The POMS-B, an emotional functioning instrument, assesses mood, tension, and other psychological symptoms and consists of 30-items assessed on a 5-point scale (0=not at all to 4=extremely). 6 summary scores are calculated: Tension/Anxiety, Depression/Rejection, Anger/Hostility, Vigor/Activity, Fatigue/Inertia, and Confusion/Bewilderment; and range from 0-20 (higher scores = more negative mood state). Analysis of this endpoint is based on the change from baseline (BL) (EOMT score minus the BL score) using an ANCOVA model with BL value, BMI, grouped center as covariates.
Time Frame: Baseline and EOMT (representing the earliest date of Week 13 visit/withdrawal visit)
Population: ITT Population. Not all participants completed a POMS-B at both Baseline and Week 13/Withdrawal; as such, the number analyzed is different from the full ITT Population counts.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | GEn 1200 mg/Day | GEn 2400 mg/Day | GEn 3600 mg/Day | PGB 300 mg/Day
Number analyzed (Participants) | 112 | 57 | 44 | 107 | 61
scores on a scale
  Tension/Anxiety Domain Score | -1.0 (0.29) | -0.6 (0.41) | -0.7 (0.47) | -0.9 (0.30) | -0.3 (0.40)
  Depression/Rejection Domain Score | -0.5 (0.30) | -0.2 (0.43) | -0.6 (0.49) | -0.3 (0.32) | 0.4 (0.41)
  Anger/Hostility Domain Score | -0.5 (0.32) | -0.8 (0.45) | -0.5 (0.51) | -0.3 (0.33) | -0.3 (0.44)
  Vigor/Activity Domain Score | 0.6 (0.32) | -0.1 (0.45) | 0.1 (0.51) | 0.7 (0.33) | -0.4 (0.44)
  Fatigue/Inertia Domain Score | -0.8 (0.37) | -0.5 (0.52) | -1.1 (0.59) | -1.1 (0.38) | -0.1 (0.50)
  Confusion/Bewilderment Domain Score | -0.3 (0.21) | 0.2 (0.29) | -0.1 (0.33) | 0.0 (0.22) | -0.2 (0.28)

ADVERSE EVENTS:
Description: Adverse events (AEs) and serious adverse events (SAEs) were captured for all participants in the Safety Population, comprised of all randomized participants who took at least one dose of investigational product.
Arm/Group | Placebo | GEn 1200 mg/Day | GEn 2400 mg/Day | GEn 3600 mg/Day | PGB 300 mg/Day
Serious Adverse Events (participants affected / at risk) | 6/120 | 3/62 | 4/56 | 5/116 | 2/66
Other Adverse Events (participants affected / at risk) | 50/120 | 34/62 | 25/56 | 62/116 | 32/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=120) | GEn 1200 mg/Day (N=62) | GEn 2400 mg/Day (N=56) | GEn 3600 mg/Day (N=116) | PGB 300 mg/Day (N=66)
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Partial seizures (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Infected skin ulcer (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Affective disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=120) | GEn 1200 mg/Day (N=62) | GEn 2400 mg/Day (N=56) | GEn 3600 mg/Day (N=116) | PGB 300 mg/Day (N=66)
Dizziness (Nervous system disorders) | 6 | 9 | 8 | 16 | 9
Somnolence (Nervous system disorders) | 5 | 2 | 7 | 14 | 9
Nausea (Gastrointestinal disorders) | 9 | 7 | 4 | 7 | 3
Oedema peripheral (General disorders) | 5 | 2 | 0 | 10 | 11
Headache (Nervous system disorders) | 9 | 3 | 4 | 4 | 6
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 6 | 0 | 11 | 3
Diarrhoea (Gastrointestinal disorders) | 6 | 3 | 2 | 6 | 5
Urinary tract infection (Infections and infestations) | 5 | 3 | 4 | 6 | 4
Constipation (Gastrointestinal disorders) | 4 | 3 | 4 | 4 | 6
Fatigue (General disorders) | 3 | 3 | 3 | 5 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 1 | 2 | 5 | 3
Nasopharyngitis (Infections and infestations) | 5 | 1 | 2 | 4 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 4 | 6 | 2
Vision blurred (Eye disorders) | 5 | 0 | 3 | 2 | 3
Weight increased (Investigations) | 1 | 0 | 2 | 5 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1 | 3 | 3
Increased appetite (Metabolism and nutrition disorders) | 4 | 0 | 3 | 1 | 3
Dry mouth (Gastrointestinal disorders) | 4 | 0 | 4 | 1 | 1
Disturbance in attention (Nervous system disorders) | 2 | 2 | 0 | 2 | 3
Vomiting (Gastrointestinal disorders) | 3 | 3 | 1 | 2 | 0
Bronchitis (Infections and infestations) | 1 | 3 | 1 | 1 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1 | 3
Hypoaesthesia (Nervous system disorders) | 1 | 1 | 1 | 0 | 3
Paraesthesia (Nervous system disorders) | 0 | 2 | 1 | 0 | 3
Fall (Injury, poisoning and procedural complications) | 0 | 3 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.